CLINICAL TRIAL: NCT06001372
Title: TREK: Ketamine-assisted Psychotherapy (KAP) for Patients With Existential Distress Associated With Non-operable GI Cancers
Brief Title: Ketamine-assisted Psychotherapy (KAP) for Patients With Existential Distress Associated With Non-operable GI Cancers
Acronym: TREK
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Challenges with feasibility
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI160227
Record Dates: First submitted 2023-08-04; First posted 2023-08-21 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Gastrointestinal Cancer; Depression; Anxiety
Keywords: Ketamine Assisted Therapy; Existential Distress
MeSH Terms: conditions — Gastrointestinal Neoplasms; Depression; Anxiety Disorders | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Single group, open label pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm 1 (Experimental): Three 2.5-3 hour Ketamine Assisted Psychotherapy sessions, each 2-7 days apart
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine, 0.5-1.2mg/kg, administered intramuscularly
  * Doses can range 0.5-1.2 mg/kg. Starting dose for all participants will be 0.5mg/kg.
  * Dose can be titrated up to maximum of 1.2 mg/kg or titrated down to 0.5 mg/kg based on response and clinical judgement.
  * Dose will be administered by injecting into large muscle mass (eg, deltoid, gluteal muscle, thigh)
  Other Names: Ketamine Assisted Psychotherapy

SUMMARY:
The goal of this open-label clinical trial is to assess the feasibility of Ketamine-assisted psychotherapy (KAP) studies for adults with non-operable GI cancers suffering with existential distress. The main questions it aims to answer are:

* Is it feasible to conduct a KAP study with this population?
* What is the safety and tolerability of KAP in this population?
* How prevalent is existential distress in this population?

Participants will undergo KAP administered as standard of care at the HMHI Park City Ketamine-Assisted Psychotherapy Clinic and will complete health assessments over the course of the study, as well as during the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged ≥ 18 years.
* Participant with non-operable GI cancers requiring multi-modal treatment (e.g. surgery +/- chemo +/-radiation) and have a a high likelihood of recurrence and/or treatment failure in the opinion of the treating investigator.
* Screen positivity for existential distress on the EDS, defined as scoring ≥ 3 on any of the 10 component domains, or a total score ≥ 6
* ECOG Performance Status ≤ 2.
* Adequate hepatic function as defined as:

  * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN) unless elevated bilirubin is related to Gilbert's Syndrome
  * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN

    * Subjects with liver metastases will be allowed to enroll with AST and ALT levels ≤ 5 x ULN.
* For participants of childbearing potential: Negative pregnancy test or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Participants < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or
    * Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Participants ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago; or
    * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Participants of childbearing potential and subjects with a sexual partner of childbearing potential must agree to use a highly effective method of contraception.
* Participants with a sexual partner of childbearing potential must agree to use a condom during intercourse for 24 hours post- ketamine dose.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, ondansetron, cannabis, and non-routine PRN medications within 24 hours of each ketamine administration. Exceptions include daily use of caffeine, nicotine, and opioid pain medication
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Agree that for one week preceding the ketamine session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the research team. Exceptions will be evaluated by the research team and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
* Agree not to use nicotine for at least 2 hours before the ketamine administration or for the duration of the ketamine session.
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the morning of the ketamine session. If the participant does not routinely consume caffeinated beverages, he or she must agree not to do so on the day of ketamine administration.
* Participants requiring opioid use for pain are on a stable pain management regimen or do not experience clinically significant sedation during opioid use. Note: Long-acting opioid medications (e.g., oxycodone sustained-release, morphine sustained release) will be allowed if the last dose occurred at least 6 hours before ketamine administration; such medication will not be taken again until at least 6 hours after ketamine administration.
* Fluent in English.
* Reading literacy and comprehension sufficient for understanding the consent form and study questionnaires, as evaluated by study staff obtaining consent.
* Have a support person who is be able to escort the participant home from the ketamine dosing sessions. Note: The use of ride services will not be permitted (e.g., Uber, Lift, taxi, etc.)

Exclusion Criteria:

* Received ketamine treatments for a psychiatric condition within 6 months of enrollment.
* Personal history or first- or second-degree relatives with schizophrenia, bipolar affective disorder, delusional disorder, schizoaffective disorder, psychosis, or other psychotic spectrum illness.
* Currently meeting DSM-5 criteria for Dissociative Disorder, or other psychiatric conditions judged to be incompatible with the establishment of rapport or safe exposure to ketamine.
* Currently meeting DSM-5 criteria for Cluster B Personality Disorder.
* Severe depression requiring immediate standard-of-care treatment (e.g., hospitalization).
* Suicidal ideation over the past month as assessed as a yes to question 3, 4, or 5 on the Columbia-Suicide Severity Rating Scale, Suicidal Ideation section
* Cancer with known CNS involvement, previously treated brain metastasis, or other major CNS disease.
* Current or history within the last two years of meeting DSM-V criteria of substance use disorder (excluding caffeine and nicotine). Current substance use disorders may be identified through the drug urine screening test.
* Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Any grade congestive heart failure, unstable angina pectoris, serious cardiac arrhythmias including tachycardia, or clinically significant screening ECG abnormalities.
    * Cardiac hypertrophy or artificial heart valve.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic events, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism), and/or significant coronary artery disease within 3 months before the first dose.
    * QTc prolongation defined as a QTcF > 450 ms.
    * Known congenital long QT.
    * Uncontrolled hypertension defined as ≥ 140/90 as assessed from the mean of three consecutive blood pressure measurements taken over 10 minutes.
  * Seizure disorder
  * Moderate to severe dementia
  * History of significant traumatic brain injury
  * Requires the use of supplemental oxygen.
  * Renal insufficiency as defined as creatinine clearance < 40 mL/min calculated by Cockcroft-Gault formula
  * Any other condition that would, in the Investigator's judgment, contraindicate the participant's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [participants may not receive the drug through a feeding tube], social/ psychological issues, etc.)
* Known HIV infection with a detectable viral load within 6 months of the anticipated start of treatment. Note: Participants on effective antiretroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), or hepatitis C. Note: Participants with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Participants positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Medical, psychiatric, cognitive, or other conditions that may compromise the participant's ability to understand the participant information, give informed consent, comply with the study protocol or complete the study.
* Known prior severe hypersensitivity to ketamine or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
* Participants taking prohibited medications as described in Section 6.5.1. A washout period of prohibited medications for a period of at least five half-lives or as clinically indicated should occur before the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Lewis, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Three 2.5-3 hour Ketamine Assisted Psychotherapy sessions, each 2-7 days apart
  Ketamine: Ketamine, 0.5-1.2mg/kg, administered intramuscularly
  * Doses can range 0.5-1.2 mg/kg. Starting dose for all participants will be 0.5mg/kg.
  * Dose can be titrated up to maximum of 1.2 mg/kg or titrated down to 0.5 mg/kg based on response and clinical judgement.
  * Dose will be administered by injecting into large muscle mass (eg, deltoid, gluteal muscle, thigh)
Period: Overall Study
Arm/Group | Arm 1
Started | 2
Completed | 1
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (15.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Study Completion by Enrolled Participants. Study Completion is Defined as Participating in at Least 2 of the 3 Ketamine-Assisted Psychotherapy (KAP) Sessions.
Description: To assess the feasibility of completion of the study intervention. This outcome measure will report the number of participants who reached study completion. Study completion was defined as participating in at least 2/3 of the 3 KAP sessions.
Time Frame: Up to 3 KAP sessions (2 weeks from the initiation of study treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 2
Participants
  Number of subjects who reached study completion. | 2
  Number of subjects who did not reach study completion. | 0

2. Secondary Outcome: The Severity of Adverse Events (AEs)
Description: This outcome will report the count of AEs and SAEs characterized by severity (as defined by the NIH CTCAE, version 5.0) to assess the safety and tolerability of ketamine-assisted therapy in the study population. All subjects who receive any study treatment will be included in the final summaries and listings of safety data. The severity of the AEs was graded according to the CTCAE v5.0. The CTCAE uses a 5-point grading system to assess the severity of AEs:
  * Grade 1: Mild
  * Grade 2: Moderate
  * Grade 3: Severe
  * Grade 4: Life-threatening
  * Grade 5: Death
  This outcome measure will report the count of participants who experienced an AE or SAE at each toxicity grade. Adverse events were followed until 14 days after the last dose of study treatment.
Time Frame: up to 48 days after initiation of the study treatment (30 days after the last dose of study treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 2
Participants
  Toxicity Grade 1: Yes | 1
  Toxicity Grade 1: No | 1
  Toxicity Grade 2: Yes | 1
  Toxicity Grade 2: No | 1
  Toxicity Grade 3: Yes | 0
  Toxicity Grade 3: No | 2
  Toxicity Grade 4: Yes | 0
  Toxicity Grade 4: No | 2
  Toxicity Grade 5: Yes | 0
  Toxicity Grade 5: No | 2

3. Secondary Outcome: To Determine the Prevalence of Existential Distress in Patients With Non-operable GI Cancers.
Description: This outcome will report the proportion of screened patients that meet Existential Distress Scale (EDS) criteria (Single domain score ≥ 3 or Total score ≥ 6). EDS is a 10-item questionnaire for subjects to rank questions about distressing thoughts from 0 to 4 (0 as not distressed, 4 as unbearably distressed). A higher score represents a higher level of Existential Distress.
  This outcome will report the count of subjects meeting EDS criteria at the following visits Ketamine Session 1, Ketamine Session 2, Ketamine Session 3, Follow-Up Day 14, Follow-Up Day 30, and Follow-Up Day 90.
Time Frame: Ketamine Session 1 (up to 1 day), Ketamine Session 2 (up to 7 days), Ketamine Session 3 (up to 15 days), Follow-Up Day 14 (up to 29 days), Follow-Up Day 30 (up to 48 days), and Follow-Up Day 90 (up to 100 days).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 2
Participants
  Ketamine Session 1: Criteria (Single domain ≥ 3 or total score ≥ 6) | 2
  Ketamine Session 1: Not Meeting Criteria (Single domain < 3 or total score < 6) | 0
  Ketamine Session 1: Not Assessed | 0
  Ketamine Session 2: Criteria (Single domain ≥ 3 or total score ≥ 6) | 2
  Ketamine Session 2: Not Meeting Criteria (Single domain < 3 or total score < 6) | 0
  Ketamine Session 2: Not Assessed | 0
  Ketamine Session 3: Criteria (Single domain ≥ 3 or total score ≥ 6) | 1
  Ketamine Session 3: Not Meeting Criteria (Single domain < 3 or total score < 6) | 0
  Ketamine Session 3: Not Assessed | 1
  Follow-Up Day 14: Criteria (Single domain ≥ 3 or total score ≥ 6) | 0
  Follow-Up Day 14: Not Meeting Criteria (Single domain < 3 or total score < 6) | 1
  Follow-Up Day 14: Not Assessed | 1
  Follow-Up Day 30: Criteria (Single domain ≥ 3 or total score ≥ 6) | 0
  Follow-Up Day 30: Not Meeting Criteria (Single domain < 3 or total score < 6) | 1
  Follow-Up Day 30: Not Assessed | 1
  Follow-Up Day 90: Criteria (Single domain ≥ 3 or total score ≥ 6) | 0
  Follow-Up Day 90: Not Meeting Criteria (Single domain < 3 or total score < 6) | 1
  Follow-Up Day 90: Not Assessed | 1

ADVERSE EVENTS:
Time Frame: AEs and SAEs were recorded from consent until 30 days after the last dose of study medication or until new cancer therapy was started, up to 48 days after initiation of study treatment.
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=2)
Suicidal ideation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=2)
Fatigue (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT06001372/Prot_SAP_000.pdf